CLINICAL TRIAL: NCT00006459
Title: Phase III Study of Gemcitabine Plus Paclitaxel Versus Paclitaxel in Patients With Unresectable, Locally Recurrent or Metastatic Breast Cancer
Brief Title: Paclitaxel With or Without Gemcitabine in Treating Women With Advanced Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Purpose: Treatment
Other Study IDs: 2017; LILLY-B9E-MC-JHQG; CDR0000068216
Record Dates: First submitted 2000-11-06; First posted 2004-02-12 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2002-04

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Paclitaxel

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known if paclitaxel is more effective with or without gemcitabine for advanced breast cancer.

PURPOSE: Randomized phase III trial to study the effectiveness of paclitaxel with or without gemcitabine in treating women who have advanced breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare overall survival of patients with unresectable, locally recurrent, or metastatic breast cancer treated with paclitaxel with or without gemcitabine.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms. Patients receive paclitaxel with or without gemcitabine. Treatment continues every 21 days in the absence of disease progression. Patients are followed every 2-4 months for 2 years after active treatment.

PROJECTED ACCRUAL: Not specified

National Cancer Institute (NCI) registered this trial with Eli Lilly as sponsor. NCI did not update the record when the trial completed. In June 2012, NCI transferred the trial to Lilly's clinicaltrials.gov account and Lilly updated the record with the trial completion date. This trial is not an applicable trial under Food and Drug Administration Amendments Act of 2007 (FDAAA).

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven unresectable, locally recurrent, or metastatic breast cancer not amenable to surgery or radiotherapy of curative intent No inflammatory breast cancer unless evidence of metastatic disease No bone metastases, pleural effusion, or ascites as the only site of disease Clinically measurable disease outside previously irradiated area Relapse after 1 prior adjuvant or neoadjuvant chemotherapy regimen containing anthracycline unless clinically contraindicated No known or suspected brain metastases or recurrence requiring steroids or radiotherapy Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Female Menopausal status: Not specified Performance status: Karnofsky 70-100% Life expectancy: At least 12 weeks Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9.0 g/dL Hepatic: ALT and AST no greater than 2 times upper limit of normal (ULN) Bilirubin no greater than 1.5 times ULN Renal: Calcium no greater than 1.2 times ULN Creatinine no greater than 1.5 times ULN Cardiovascular: No active uncontrolled cardiac disease and/or myocardial infarction within the past 6 months Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 3 months after completion of study No other prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix No other serious systemic disorder precluding study No active infection No severe psychiatric disease No history of hypersensitivity reactions to polyoxyethylated castor oil-based drugs

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior bone marrow transplantation or autologous stem cell infusion following high-dose adjuvant chemotherapy for metastatic disease No concurrent immunotherapy (including humanized anti-HER2 antibody) Chemotherapy: See Disease Characteristics See Biologic therapy No prior chemotherapy for metastatic breast cancer No prior gemcitabine or taxane No other concurrent chemotherapy Endocrine therapy: See Disease Characteristics Prior antitumoral hormonal therapy allowed No concurrent hormonal therapy excluding contraceptives and replacement steroids Radiotherapy: See Disease Characteristics At least 2 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: See Disease Characteristics Other: Recovered from prior therapy At least 30 days since prior investigational drugs No concurrent investigational drugs Concurrent bisphosphonate therapy allowed if not begun or stopped within 4 weeks before study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-07; Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Furhan Yunus, MD, FACP, Study Chair — University of Tennessee
Locations (31):
- United States (31):
  - Comprehensive Cancer Institute of Huntsville, Huntsville, Alabama
  - Little Rock Hematology-Oncology Associates, Little Rock, Arkansas
  - Pacific Coast Hematology/Oncology Medical Group, Fountain Valley, California
  - Office of Alex J.P. Makalinao, Los Angeles, California
  - Hematology/Oncology Group, Santa Rosa, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Danbury Internal Medicine, Danbury, Connecticut
  - Comprehensive Cancer Care Specialists of Boca Raton, Boca Raton, Florida
  - Mercy Hospital, Miami, Florida
  - Mountain States Tumor Institute, Boise, Idaho
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Indiana Community Cancer Care, Inc., Indianapolis, Indiana
  - Cancer Health Associates, Michigan City, Indiana
  - North Mississippi Hematology and Oncology Associates, Ltd., Tupelo, Mississippi
  - St. John's Mercy Medical Center, St Louis, Missouri
  - APN-IMPATH Research Corporation, Fort Lee, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - HemOnCare, P.C., Brooklyn, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - N.W. Carolina Oncology & Hematology, P.A., Hickory, North Carolina
  - Oklahoma Oncology Inc., Tulsa, Oklahoma
  - Rittenhouse Hematology/Oncology, Philadelphia, Pennsylvania
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Office Of C. Michael Jones, Germantown, Tennessee
  - Boston Baskin Cancer Group, University Tennessee Oncology/Hematology Group, Memphis, Tennessee
  - University of Tennessee, Memphis, Memphis, Tennessee
  - Arlington Cancer Center, Arlington, Texas
  - Southwest Regional Cancer Center, Austin, Texas
  - Intermountain Hematology/Oncology Associates, Inc., Salt Lake City, Utah
  - Northern Virginia Oncology Group, P.C., Fairfax, Virginia

REFERENCES:
- [Derived] Smyth EN, Shen W, Bowman L, Peterson P, John W, Melemed A, Liepa AM. Patient-reported pain and other quality of life domains as prognostic factors for survival in a phase III clinical trial of patients with advanced breast cancer. Health Qual Life Outcomes. 2016 Mar 25;14:52. doi: 10.1186/s12955-016-0449-z. PMID 27016084